CLINICAL TRIAL: NCT02942940
Title: Conventional Follow-up Versus Mobile App Home Monitoring For Post-Operative Anterior Cruciate Ligament (ACL) Reconstruction Patients: A Randomized Controlled Trial
Brief Title: Conventional Follow-up Versus Mobile App For Post-Operative ACL Reconstruction Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto Orthopaedic Sports Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MobileApp
Record Dates: First submitted 2016-10-06; First posted 2016-10-24 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Anterior Cruciate Ligament (ACL) Tear
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mobile app (Active Comparator)
  Interventions: Device: mobile app
- in-person (Active Comparator)
  Interventions: Other: conventional in-person

INTERVENTIONS:
Device: mobile app — The mobile app follow-up group will have no planned in-person follow-up, however these visits will be replaced with surgical site examination via submitted photos, Visual Analogue Scale (VAS), and Quality of Recovery - 9 questionnaire (QoR-9) and limb specific recovery monitoring. All information is submitted with the mobile app (QoC Health Inc, Toronto).
  Arms: mobile app
Other: conventional in-person — Patients in the conventional follow-up group will have a planned clinic follow-up at 2 and 6 weeks post-operatively, which is the schedule currently used by our surgeons. At these scheduled follow-up visits, patients will be asked to complete the VAS to assess pain and the QoR-9 in addition to recovery questions about their operated extremity.
  Arms: in-person

SUMMARY:
Background: Telemedicine is increasingly used to overcome distance between patients and physicians. Preliminary studies suggest that mobile app follow-up care for ACL reconstruction patients is feasible, can avert in-person follow-up care, and is cost-effective.

Objective: To avert in-person follow-up through the use of a mobile app in the first six weeks after surgery.

Methods: This will be a single-center, prospective randomized controlled trial

Results: Data to be analyzed from 72 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing ACL reconstruction at Women's College Hospital (WCH), between the ages of 18-70.
* Patients must be able to use a mobile device and communicate in English.

Exclusion Criteria:

* Patients who are smokers, as they carry increased rates of complications.
* Patients must not:

  * Suffer from chronic pain
  * Be taking narcotic (morphine-like) medication for pain on a regular basis, and
  * Have an allergy to local anesthetics or morphine-like medications

    * Pain scores captured in the VAS and QoR-9 are important for judging post-operative recovery. Pre-existing pain or inability to take narcotics post-operatively would compromise the reliability of these measures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Required physician visits | 6 weeks post surgery
  Total number of physician visits (including specialist, family physician, and ER) related to surgery

SECONDARY OUTCOMES:
Health care phone calls | 6 weeks post surgery
  Total number of health care telephone calls and emails (including specialist, family physician and ER)

OTHER OUTCOMES:
Cost of treatment | through study completion (approximately one year)
  cost of treatment related to surgery (i.e. rehabilitation, assistive devices)
Patient satisfaction with post-operative care | 6 weeks post surgery
  patient satisfaction as recorded in the questionnaires (VAS) at 6 weeks post surgery
Patient satisfaction with post-operative care | 6 weeks post surgery
  patient satisfaction as recorded in the questionnaires (QoR-9) at 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided